CLINICAL TRIAL: NCT06292585
Title: Acute EpiDural Hematoma Treated With Middle Meningeal Artery Embolization: a Randomized Trial (AEDH-MT)
Acronym: AEDH-MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEDH-MT
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: EpiDural Hematoma; Traumatic Brain Injury
Keywords: AEDH; EDH
MeSH Terms: conditions — Hematoma, Epidural, Spinal; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): MMA embolization
  Interventions: Procedure: MMA embolization plus medical therapy
- Control group (Active Comparator): Conservative treatment
  Interventions: Drug: Medical therapy alone

INTERVENTIONS:
Procedure: MMA embolization plus medical therapy — Patients assigned to the intervention group will receive endovascular embolization treatment within 2 hours after enrollment. Patients will receive the best conservative treatment recommended by the guidelines after MMA, and conservative treatment will be the same in both groups
  Arms: Intervention group
Drug: Medical therapy alone — Patients will receive the best conservative treatment recommended by the guidelines, and conservative treatment will be the same in both groups. Conservative treatment includes medication and general treatment. Drug therapy can be divided into hemostatic treatment, antihypertensive treatment, and symptomatic treatment. Specific local clinical diagnosis and treatment standards shall prevail or refer to corresponding clinical guidelines.
  Arms: Control group

SUMMARY:
A prospective, multicenter, randomized controlled, open-label, blinded endpoint evaluation study.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled, open-label, blinded endpoint evaluation study.

All patients diagnosed with acute epidural hematoma through cranial CT will undergo neurological examination and measurement of hematoma size. For patients who meet the inclusion criteria, they will be randomly assigned 1:1 to the middle meningeal artery embolization group (intervention group) and the conservative treatment group (control group). A total of 194 subjects need to be enrolled, including 97 in the intervention group and 97 in the control group.

Primary Outcome： The proportion of patients who require craniotomy due to the progression of epidural hematoma 7 days after injury*, and neurogenic death 28 days after injury.

*This includes patients who have actually undergone surgery and those who were deemed necessary by the committee but did not undergo surgery for various reasons.

Secondary outcome：

1. Changes in hematoma volume 7±2 days after injury (or at discharge)
2. GCS score at 7±2 days after injury (or at discharge)；
3. Hematoma volume 28±7 days after injury
4. GCS score at 28±2 days after injury；
5. ICU hospitalization days；
6. Total hospitalization days;
7. Discharge rehabilitation destination (home vs rehabilitation hospital)
8. Number of re-hospitalizations；
9. GOSE score at 3 months after injury
10. EQ-5D scale scores at 3 months after injury；
11. GOSE score at 6 months after injury
12. EQ-5D scale scores at 6 months after injury

Safety outcome:

1. Perioperative surgical complications (including craniotomy and neurovascular)
2. All-cause mortality rate at 28 ± 7 days after injury;
3. All-cause mortality rate at 3 months after injury;
4. Serious adverse events (SAEs) 3 months after injury;
5. All-cause mortality rate at 6 months after injury;
6. Serious adverse events (SAEs) 6 months after injury.

ELIGIBILITY:
Inclusion Criteria：

1. Age 18 or above；
2. Patients with a clear history of head trauma and confirmed acute epidural hematoma by head CT；
3. Cases that the case screening committee deems suitable for conservative treatment*；
4. Randomly within 6 hours after injury, and initiate treatment within 8 hours after injury；
5. Epidural hematoma located on the convex surface of the brain (frontal, temporal, parietal, or occipital)；
6. The patient or their representative agrees and signs an informed consent form. * The case screening committee is composed of three senior neurosurgeons, with two of them jointly deciding whether conservative treatment is possible. If there is a disagreement, the third doctor will make the final judgment. Including but not limited to the following two situations: 1. Hematoma volume<30ml, hematoma thickness<15mm, midline shift (MLS) <5mm, GCS score>8, and no focal neurological deficit; 2. If the GCS score is ≥ 13, the imaging standards can be appropriately relaxed.

Exclusion criteria：

1. Patients who require craniotomy surgery to remove hematoma；
2. Bilateral acute epidural hematoma；
3. Combined severe acute subdural hematoma；
4. Brainstem injury；
5. There are obvious brain contusions, lacerations, intracerebral hematomas, etc；
6. Combined intracranial tumors and other intracranial space occupying diseases；
7. Severe damage to combined extracranial organs；
8. mRS score > 2 before injury；
9. Coagulation dysfunction (preoperative INR>1.5), abnormal platelet count and function (platelet < 80×109/L)；
10. There are contraindications for cerebral angiography, such as iodine contrast agent allergy, embolization material allergy etc.；
11. There may be anatomical variations that may affect the safety of MMA embolization surgery and are not suitable for endovascular embolization；
12. Severe comorbidities, may prevent improvement of the condition or completion of follow-up；
13. Having undergone major surgical procedures within 30 days before surgery；
14. Currently participating in other clinical trials；
15. Pregnant women；
16. Suffering from malignant tumors with an expected lifespan of less than 1 year；
17. Unable to complete follow-up as required by the protocol；
18. The physician believes that the patient has other circumstances that are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who require craniotomy due to the progression of epidural hematoma 7 days after injury*, and neurogenic death 28 days after injury | Within 28 days after injury
  *This includes patients who have actually undergone surgery and those who were deemed necessary by the committee but did not undergo surgery for various reasons.

SECONDARY OUTCOMES:
Changes in hematoma volume 7±2 days after injury (or at discharge) | 7±2 days after injury (or at discharge)
GCS score at 7±2 days after injury (or at discharge) | 7±2 days after injury (or at discharge)
Hematoma volume 28±7 days after injury | 28±7 days after injury
GCS score at 28±2 days after injury | 28±2 days after injury
ICU hospitalization days | 28±2 days after injury
Total hospitalization days | 28±2 days after injury
Discharge rehabilitation destination (home vs rehabilitation hospital) | 28±2 days after injury
Number of re-hospitalizations | 6 months after injury
GOSE score at 3 months after injury | 3 months after injury
EQ-5D scale scores at 3 months after injury | 3 months after injury
GOSE score at 6 months after injury | 6 months after injury
EQ-5D scale scores at 6 months after injury | 6 months after injury

OTHER OUTCOMES:
Perioperative surgical complications (including craniotomy and neurovascular) | Perioperative period
All-cause mortality rate at 28 ± 7 days after injury | 28 ± 7 days after injury
All-cause mortality rate at 3 months after injury | 3 months after injury
Serious adverse events (SAEs) 3 months after injury | 3 months after injury
All-cause mortality rate at 6 months after injury | 6 months after injury

CONTACTS AND LOCATIONS:
Overall Officials: Jianimin Liu, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to Oriental Collaboration group on Emerging Advanced therapy for Neurovascular diseases Consortium.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: http://www.ocin.org.cn/about